CLINICAL TRIAL: NCT05222412
Title: Managed Access Programs for LNP023, Iptacopan
Status: Available | Type: Expanded Access
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Other Study IDs: CLNP023B12004M
Record Dates: First submitted 2022-01-18; First posted 2022-02-03 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-12

CONDITIONS: C3 Glomerulopathy (C3G); Paroxysmal Nocturnal Hemoglobinuria (PNH)
Keywords: C3 glomerulopathy (C3G); Paroxysmal nocturnal hemoglobinuria (PNH); MAP; Manage access program; Iptacopan; LNP023
MeSH Terms: conditions — Hemoglobinuria, Paroxysmal | interventions — iptacopan

STUDY DESIGN:
Expanded Access Types: Intermediate

INTERVENTIONS:
Drug: Iptacopan — Patients receive Iptacopan
  Other Names: LNP023

SUMMARY:
The purpose of this registration form is to list all Managed Access Programs (MAPs) related to LNP023, Iptacopan

DETAILED DESCRIPTION:
* CLNP023B12004M - Available - Managed Access Program (MAP) Cohort Treatment Plan CLNP023B12004M to Provide Access to Iptacopan (LNP023) for Complement 3 Glomerulopathy in Native and Transplanted Kidneys.
* CLNP023N12001M - Available - Managed Access Program (MAP) Cohort Treatment Plan CLNP023N12001M to provide access to Iptacopan for patients with paroxysmal nocturnal hemoglobinuria (PNH).

ELIGIBILITY:
Inclusion Criteria:

* An independent request should be received from a licensed physician (in some instances from Health Authorities, Institutions or Governments).
* The patient has a serious or life-threatening disease or condition and no comparable or satisfactory alternative therapy is available for diagnosis, monitoring or treatment; patient is not medically eligible for available treatment alternatives or has exhausted all available treatment options.
* The patient is not eligible or able to enroll in a Novartis clinical trial or continue participation in a Novartis clinical trial.
* There is a potential patient benefit to justify the potential risk of the treatment use, and the potential risk is not unreasonable in the context of the disease or condition to be treated.
* The patient must meet any other medical criteria established by the medical experts responsible for the product or by the Health Authority in a country (as applicable).
* Provision of the product will not interfere with the initiation, conduct or completion of a Novartis clinical trial or overall development program.
* Managed access provision is allowed per local laws/regulations.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult